CLINICAL TRIAL: NCT02833935
Title: Pilot Randomized Controlled Trial Evaluating a Self-Determination Theory Tele-rehabilitation Physical Activity Intervention to Enhance Motivation, Physical Activity, and Quality of Life-related Outcomes Among Adults With SCI
Brief Title: Enhancing Quality of Life Through Exercise: A Tele-Rehabilitation Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Craig H. Neilsen Foundation (Other)
Collaborators: McGill University (Other)
Responsible Party: Principal Investigator, Dr. Shane Sweet, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CraigHNF
Record Dates: First submitted 2016-07-08; First posted 2016-07-14 (Estimated); Results first posted 2022-01-26 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; physical activity; self-determination theory; life satisfaction
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity; Personal Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Activity Intervention Group (Experimental): Participants will complete a baseline questionnaire (week 1) about their demographic information, self-determination theory variables, their current physical activity, and other psychological indicators. They will complete the same questionnaire at two additional time points. First, about halfway through the intervention (week 6), and then at the end (week 10). Participants in the physical activity intervention group will also receive 8 1-hour physical activity sessions over 2 months (1/week) with a trained physical activity counselor through a video-based internet platform.
  Interventions: Behavioral: Physical Activity Intervention
- Control Group (No Intervention): Control Group: For participants assigned to the control group, they will be asked to continue with their regular routine for the next two months. Otherwise, the participants in this group will be asked to complete the follow-up baseline questionnaires at 6 and 10 weeks post-baseline. They will be contacted by a physical activity counsellor at the end of the 10-week period.

INTERVENTIONS:
Behavioral: Physical Activity Intervention — The PA intervention will be delivered in a virtual face-to-face format using the secure and confidential "Remote Education, Augmented Communication, Training and Supervision" online video-based software. Intervention participants will receive 8 PA sessions over 2 months (1/week), following collaborator specific telephone-based PA counselling protocol. The counsellor will individually tailor her approach to each participant by understanding the participant's past and current PA experiences, motives to be physically active, salient concerns and barriers regarding PA, and physical home environment. Throughout the intervention, the PA counsellor and participants will co-construct and collaboratively adapt the intervention with the participants.
  Arms: Physical Activity Intervention Group

SUMMARY:
Pilot randomized controlled trial evaluating a Self-Determination Theory (SDT) video-based tele-rehabilitation physical activity intervention aimed to enhance basic psychological needs, motivation, physical activity (PA), and quality of life- related outcomes of adults with spinal cord injury (SCI). It is anticipated that the individuals who receive the physical activity intervention (intervention group) will have moderate increases in their basic psychological needs, autonomous motivation, life satisfaction, and physical activity participation, and a moderate decrease in controlled motivation and depressive symptoms compared to the individuals who did not receive the intervention (control group).

DETAILED DESCRIPTION:
Adults with spinal cord injury (SCI) report lower levels of quality of life (e.g., low life satisfaction; high depression) than the general population and have low rates of community participation. One health behavior that can improve these psychosocial outcomes is physical activity (PA). Unfortunately, PA rates are very low among adults with SCI. Novel interventions to increase PA are needed. One approach that has gained traction is video-based tele-rehabilitation, which has the benefit of reducing costs, increasing accessibility to services and delivering and adapting the intervention to the person's home environment.

Experts have strongly recommended that PA interventions be based in psychological theory to enhance their effectiveness. The intervention will be grounded in a strong psychological/motivational theory called self-determination theory (SDT). According to SDT, humans strive for growth and well-being by aiming to satisfy their three basic psychological needs of autonomy (sense of volition), competence (sense of capability) and relatedness (sense of connectedness). The investigators intervention will therefore be designed to foster these psychological needs in order to increase intrinsic/autonomous motivation for PA, promote higher PA levels and improve quality of life and participation.

To date, no study has either conducted a video-based tele-rehabilitation intervention to promote PA or has tested SDT among adults with SCI; thus providing the need for a pilot intervention. The purpose of this study is to pilot test an innovative, theory-informed, video-based tele-rehabilitation intervention aimed to enhance SDT-variables, PA and quality of life-related variables among adults with SCI. Effect sizes derived from this pilot intervention will be used to inform the sample size calculation of a subsequent larger randomized controlled trial. Given previous video-based PA tele-rehabilitation interventions do not exist, the hypotheses are derived from PA and general telephone-based counselling studies. Specifically, it is hypothesized that the video-based intervention will have moderate effects on SDT variables, PA, participation, life satisfaction and depression.

ELIGIBILITY:
Inclusion Criteria:

* Must have spinal cord injury (paraplegia)
* Must use a mobility device
* Must have sustained their injury at least 1 year prior
* Have a computer that matches requirements to use the online video-based software
* Speak and understand English or French
* Must have the intention to become physically active in the next two months or have been minimally active (< 2 times a week) in the past two months

Exclusion Criteria:

* Receiving in-patient rehabilitation services
* Have been diagnosed with memory impairments
* Have severe communication difficulties and/or severe visual impairments
* Do not require a mobility device (e.g., wheelchair, cane)
* Have answered yes to one of the questions on the Physical Activity Readiness Questionnaire (PAR-Q+) and do not have a doctor's note saying it is safe for them to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shane Sweet, PhD, Principal Investigator — McGill University
Locations (1):
- McGill University; Dept. of Kinesiology & Physical Education; Theories and Interventions in Exercise and Health Psychology Laboratory, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be shared among co-investigators.

REFERENCES:
- [Derived] Sweet SN, Rocchi M, Arbour-Nicitopoulos K, Kairy D, Fillion B. A Telerehabilitation Approach to Enhance Quality of Life Through Exercise Among Adults With Paraplegia: Study Protocol. JMIR Res Protoc. 2017 Oct 19;6(10):e202. doi: 10.2196/resprot.8047. PMID 29051134

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Physical Activity Intervention Group | Control Group
Started | 12 | 12
Completed | 10 | 12
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Physical Activity Intervention Group: Participants will complete a baseline questionnaire (week 1) about their demographic information, self-determination theory variables, their current physical activity, and other psychological indicators. They will complete the same questionnaire at two additional time points. First, about halfway through the intervention (week 6), and then at the end (week 10). Participants in the physical activity intervention group will also receive 8 1-hour physical activity sessions over 2 months (1/week) with a trained physical activity counselor through a video-based internet platform.
  Physical Activity Intervention: The PA intervention will be delivered in a virtual face-to-face format using the secure and confidential "Remote Education, Augmented Communication, Training and Supervision" online video-based software. Intervention participants will receive 8 PA sessions over 2 months (1/week), following collaborator specific telephone-based PA counselling protocol.
- Total: Total of all reporting groups
Arm/Group | Physical Activity Intervention Group | Control Group | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.64 (12.64) | 53 (11.29) | 50.50 (12.34)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One missing data
  Participants
    number analyzed (Participants) | 11 | 12 | 23
    Female | 5 | 2 | 7
    Male | 6 | 10 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 12 | 11 | 23
  Race: Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 11 | 10 | 21
  United States | 1 | 2 | 3
Mobility Mode [Count of Participants; unit: Participants] — Missing data Population: Missing data
  Participants
    number analyzed (Participants) | 11 | 11 | 22
    Manual Wheelchair | 8 | 7 | 15
    Other (e.g., cane) | 3 | 4 | 7
Cause of Spinal Cord Injury [Count of Participants; unit: Participants]
  Traumatic | 8 | 8 | 16
  Non-Traumatic | 4 | 4 | 8
Language [Count of Participants; unit: Participants]
  Francophone | 8 | 9 | 17
  Anglophone | 4 | 3 | 7
Years since Spinal Cord Injury [Mean (Standard Deviation); unit: years] | 15.8 (14.51) | 15.10 (10.89) | 15.45 (12.85)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Self-Regulation for Exercise Scale
Description: Measure to assess changes in autonomous and controlled types of motivation for reasons why one would exercise/engage in physical activity throughout the intervention. A total scale score range of 1 (not at all true) to 7 (very true) will be used to respond to 15 items. A mean score of participants' autonomous (6 items; " Because I personally believe it is the best thing for my health.") and controlled motivation (6 items; "Because I want others to approve of me.") will be calculated. A higher value indicates greater autonomous and or controlled types of motivation.
Time Frame: Baseline, Week 6, and Week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Activity Intervention Group | Control Group
Number analyzed (Participants) | 10 | 12
score on a scale
  Autonomous Motivation (Baseline) | 5.75 (1.50) | 5.51 (1.15)
  Controlled Motivation (Baseline) | 3.23 (1.40) | 2.63 (0.89)
  Autonomous Motivation (6 weeks) | 6.33 (0.75) | 5.63 (0.98)
  Controlled Motivation (6 weeks) | 2.55 (1.17) | 2.79 (0.88)
  Autonomous Motivation (10 weeks) | 6.32 (0.97) | 5.31 (1.21)
  Controlled Motivation (10 weeks) | 2.65 (0.97) | 2.63 (0.80)

2. Primary Outcome: Psychological Needs for Exercise Questionnaire
Description: Measure to assess changes during the intervention in the basic psychological needs for exercise as per self-determination theory. Data will be collected at baseline, week 6, and week 10 for both participant groups. On a 6-point likert scale ranging from 1 (false) to 6 (true), participants will respond to 18 items reflecting how they might feel when physically active. After summating all items, a total mean score was calculated for autonomy (6 items; "I feel free to exercise in my own way"), competence (6 items; "I feel that I am able to complete exercises that are personally challenging"), and relatedness (6 items; "I feel close to my exercise companions who appreciate how difficult exercise can be"). A higher value indicates greater need satisfaction. Total values are reported in the data table as a sum of all 3 categories (Score range is 3-18).
Time Frame: Baseline, Week 6, and Week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Activity Intervention Group | Control Group
Number analyzed (Participants) | 10 | 12
score on a scale
  Baseline | 4.52 (0.84) | 4.50 (1.03)
  6 weeks | 4.36 (0.96) | 4.61 (0.70)
  10 weeks | 4.51 (0.96) | 4.43 (0.74)

3. Secondary Outcome: Leisure Time Physical Activity Questionnaire for People With Spinal Cord Injury
Description: Questionnaire used to measure physical activity levels. Participants will be asked to indicate the frequency (days) and duration (in minutes) they engage in mild, moderate, and vigorous intensity activities over the last 7 days. Weekly minutes of total activity (mild, moderate, and vigorous) and of moderate and vigorous activity will be summed.
Time Frame: Baseline, Week 6, and Week 10
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Physical Activity Intervention Group | Control Group
Number analyzed (Participants) | 10 | 12
Minutes
  Total (Baseline) | 116.70 (175.54) | 114.17 (208.82)
  Total (6 weeks) | 375.82 (334.12) | 149.30 (194.75)
  Total (10 weeks) | 505.82 (322.84) | 253.36 (272.15)

4. Secondary Outcome: Person-Perceived Participation in Daily Activities Questionnaire
Description: Measure to assess participation in daily and social activities. Participants will be presented with a list of 26 activities. For each activity, they are asked, "Do you participate in this activity?" Response options are "Yes, as much as I want" (4); "Yes, but less than I want"(3); "No, but I would like to" (2); and "No, but I don't want to" (1). An overall participation in daily and social activities score will be calculated as well as six sub-scale scores reflecting broad categories of participation will be summed. The 6 subscales are autonomous participation- indoors (7 items, range 7-28), autonomous participation-outdoors (6 items, range 6-24), family roles (4 items, range 4-16), health (2 items, range 2-8), social relationships (4 items, range 4-16), work-education (3 items, range 3-12). Each sub-scale is calculated by adding the scores of the individual items. A higher score of each category indicates greater participation.
Time Frame: Baseline, Week 6, and Week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Activity Intervention Group | Control Group
Number analyzed (Participants) | 10 | 12
score on a scale
  Health Participation (baseline) | 4.30 (1.06) | 4.50 (1.17)
  Health Participation (6 weeks) | 5.20 (0.92) | 4.09 (1.30)
  Health Participation (10 weeks) | 5.10 (0.99) | 4.09 (3.02)
  autonomous participation- indoors (baseline) | 19.6 (1.51) | 18.67 (3.89)
  autonomous participation- indoors (6 weeks) | 19.4 (1.84) | 19.72 (1.68)
  autonomous participation- indoors (10 weeks) | 19.9 (0.88) | 18.18 (3.31)
  autonomous participation-outdoors (baseline) | 12.2 (4.13) | 14 (3.41)
  autonomous participation-outdoors (6 weeks) | 11.5 (3.60) | 14.36 (2.58)
  autonomous participation-outdoors (10 weeks) | 13.1 (3.38) | 13.27 (2.76)
  family roles (baseline) | 9.5 (1.84) | 8.92 (2.87)
  family roles (6 weeks) | 9.7 (1.57) | 10 (1.61)
  family roles (10 weeks) | 9.3 (0.82) | 8.55 (2.42)
  social relationships (baseline) | 11 (0.82) | 10.5 (2.39)
  social relationships (6 weeks) | 10.8 (1.14) | 10.63 (1.21)
  social relationships (10 weeks) | 10.7 (1.95) | 10.36 (1.43)
  work-education (baseline) | 3.8 (3.46) | 5.58 (2.78)
  work-education (6 weeks) | 3.6 (3.31) | 6.45 (2.16)
  work-education (10 weeks) | 4.2 (3.68) | 4.91 (3.02)

5. Secondary Outcome: Life Satisfaction Questionnaire
Description: Standardized and validated quality of life measure that asks 11 questions about satisfaction in various areas of life, including life in general, vocation, financial situation, leisure, social/friends/family, sexual life, family life, and physical and mental health (1=very dissatisfying to 6=very satisfying). The mean score of the 11 items will be calculated for this measure.
Time Frame: Baseline, Week 6, and Week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Activity Intervention Group | Control Group
Number analyzed (Participants) | 10 | 12
score on a scale
  Baseline | 4.41 (0.76) | 4.31 (0.92)
  6 weeks | 4.42 (0.75) | 4.17 (0.95)
  10 weeks | 4.64 (0.70) | 4.23 (0.89)

6. Secondary Outcome: Patient Health Questionnaire
Description: Measures symptoms of depression using 9 items. Participants will be asked, "Over the past 4 weeks, how often have you been bothered by any of the following problems?" and rate each symptom (eg, little interest or pleasure in doing things, poor appetite or overeating) on a 4-point scale (0=not at all; 1=Several days; 2=More than half the days 3=nearly every day). A mean score of the items will be computed with higher scores indicating higher reported symptoms of depression.
Time Frame: Baseline, Week 6, and Week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Activity Intervention Group | Control Group
Number analyzed (Participants) | 10 | 12
score on a scale
  Baseline | 0.50 (0.44) | 0.56 (0.62)
  6 weeks | 0.56 (0.41) | 0.68 (0.66)
  10 weeks | 0.63 (0.44) | 0.56 (0.62)

7. Secondary Outcome: Health Care Climate Questionnaire
Description: Measures self-determination theory perspective on need support. Participants will respond to six items (e.g., "My exercise counselor listened to how I would like to do things regarding my exercise") on a 7-point Likert scale ranging from strongly disagree (1) to strongly agree (7). A higher mean score indicates greater perceptions of need support.
Time Frame: Baseline, Week 6, and Week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Activity Intervention Group
Number analyzed (Participants) | 10
score on a scale
  Baseline | 6.55 (.43)
  Week 6 | 6.67 (.49)
  Week 10 | 4.13 (.49)

8. Other Pre Specified Outcome: Positive Affect and Negative Affect Schedule Questionnaire
Description: A measure of affective experience capturing broader aspects of well-being/quality of life
Time Frame: Baseline, Week 6, and Week 10
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Meaning Questionnaire
Description: Measures meaningful life experience capturing broader aspects of well-being/quality of life. This 5-item scale asks participants to rate their responses from 1 (absolutely untrue) to 7 (absolutely true). A higher score indicated greater reported meaning.
Time Frame: Baseline, Week 6, and Week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Activity Intervention Group | Control Group
Number analyzed (Participants) | 10 | 12
score on a scale
  Baseline | 5.40 (1.53) | 5.11 (1.42)
  6 weeks | 5.30 (0.87) | 5.02 (1.08)
  10 weeks | 5.50 (0.95) | 4.78 (1.03)

10. Other Pre Specified Outcome: Social Cognitive Predictors of Leisure Time Physical Activity (LTPA) Among Adults With Spinal Cord Injury (e.g., Self-efficacy, Intentions, Action Planning)
Description: This measure consists of a battery of short questionnaires assessing psychosocial predictors of leisure time exercise activity such as self-efficacy, intentions, and action planning among adults with spinal cord injury. Intentions were measured with 2 items and participants responded on a scale (1-strongly disagree 7-strongly agree). Action planning was measured with 4 items and participants responded on a scale (1-definitely false 7-definitely true). Barrier self efficacy was measured with 6 items and task efficacy was measured with 8 items and participants responded on a scale (1-not at all confident 7-completely confident). A higher score on each of the questionnaires indicated higher levels (e.g., greater intentions, self-efficacy, and action planning).
Time Frame: Baseline, Week 6, and Week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Activity Intervention Group | Control Group
Number analyzed (Participants) | 10 | 12
score on a scale
  Intentions (baseline) | 4.70 (2.20) | 4.58 (1.96)
  Intentions (6 weeks) | 5.50 (1.16) | 4.66 (1.84)
  Intentions (10 weeks) | 5.05 (2.43) | 4.33 (1.37)
  Barrier self-efficacy (baseline) | 5.42 (1.36) | 4.65 (1.57)
  Barrier self-efficacy (6 weeks) | 5.00 (1.60) | 3.98 (1.41)
  Barrier self-efficacy (10 weeks) | 5.17 (1.14) | 3.94 (1.20)
  Action planning (baseline) | 5.40 (1.36) | 4.48 (1.62)
  Action planning (6 weeks) | 5.54 (1.81) | 4.02 (2.16)
  Action planning (10 weeks) | 5.45 (1.31) | 4.10 (2.07)

11. Other Pre Specified Outcome: Behavioural Regulation in Exercise Questionnaire
Description: Measure to assess changes in all 6 motivational regulations as per self-determination theory asking reasons why individuals engage in exercise/physical activity during the intervention. Participants will respond to 23 items (e.g, "I don't see why I should have to exercise"), on a 5-point Likert scale ranging from 0 (not true for me) to 4 (very true for me), covering the types of motivational regulations on the self-determination continuum. The mean score of participants' autonomous and controlled motivation will be calculated. A higher mean score indicated a higher level of that type of motivation. Outcome measure data are not presented because of missingness.
Time Frame: Baseline, Week 6, and Week 10
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not assessed.
Arm/Group | Physical Activity Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT02833935/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT02833935/SAP_001.pdf